CLINICAL TRIAL: NCT02560194
Title: Evaluation of Flexible Sigmoidoscopy Screening as an Adjunct to the National FOBT Screening Programme in Scotland - A Random Evaluation
Brief Title: Evaluation of Flexible Sigmoidoscopy Screening as an Adjunct to the National FOBT Screening Programme in Scotland
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Dundee (Other)
Responsible Party: Principal Investigator, Professor Robert J C Steele, Professor of Surgery, University of Dundee
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2013ON22
Record Dates: First submitted 2015-09-03; First posted 2015-09-25 (Estimated); Last update posted 2018-03-23 (Actual); Status verified 2018-03

CONDITIONS: Colorectal Cancer; Colorectal Adenoma
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Occult Blood

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Flexible Sigmoidoscopy (Active Comparator): People randomized to this arm are offered flexible sigmoidoscopy in addition to FOBT at the age of 60.
  Interventions: Procedure: Flexible Sigmoidoscopy
- FOBT only (Placebo Comparator): People in this are offered fecal occult blood testing only.
  Interventions: Other: Fecal occult blood test

INTERVENTIONS:
Procedure: Flexible Sigmoidoscopy — Examination of the rectal and distal colon by means of a flexible endoscope
  Arms: Flexible Sigmoidoscopy
Other: Fecal occult blood test — Test for hemoglobin in faeces
  Arms: FOBT only

SUMMARY:
Guaiac faecal occult blood testing (gFOBT) consistently demonstrates reductions in deaths from colorectal cancer of around 16% and gFOBT screening is now routine in all four countries of the United Kingdom. However, gFOBT has significant limitations and is associated with a substantial interval cancer rate in the region of 50 %, indicating a severe deficiency in sensitivity for cancer. Additionally, as the majority of colorectal cancers arise from pre-existing adenomas, it is important for colorectal screening programmes to detect adenomas in order to reduce the incidence of the disease as well as the associated mortality. Although gFOBT does detect some adenomas, most randomised trials have not demonstrated a reduction in colorectal cancer incidence. Also, FOBT screening tends to under-detect cancers in women and it is relatively insensitive for rectal cancer when compared with colon cancer.

Single flexible sigmoidoscopy (FS), between the ages of 55 and 65 years, has been shown to bring about a significant reduction in colorectal cancer mortality. In addition, and most importantly, after a period of four years a significant reduction in colorectal cancer incidence was observed. FS does not suffer from low specificity since false positives do not occur, and there is independent evidence that it is more sensitive than a single gFOBT. In addition, FS is ideally suited to detecting rectal cancers and adenomas, and it is unlikely that there would be a gender difference in the sensitivity.

Single FS has not been compared with biennial FOBT and there is no information regarding the utility of FS in a population that has already been exposed to FOBT screening. It is hypothesised that offering a combination of gFOBT and FS would provide an enhanced screening algorithm that would be associated with better outcomes than gFOBT alone. In order to test this hypothesis a randomised evaluation pilot study of FS screening integrated into the current gFOBT Screening Programme, will be carried out in those around age 60, as this appears to be the age at which adenoma prevalence peaks.

DETAILED DESCRIPTION:
Screening for colorectal cancer is now being introduced in many countries worldwide, but there is still considerable uncertainty as to the ideal modality. Population based trials of guaiac faecal occult blood testing (gFOBT) have consistently demonstrated significant reductions in disease specific mortalities and three randomised population based trials of biennial gFOBT have demonstrated reductions in deaths from colorectal cancer of around 16%. As a result of these trials, a demonstration pilot was performed in the United Kingdom which has led to the introduction of gFOBT screening in all four countries of the United Kingdom.

However, gFOBT has significant limitations. It is clear that this form of screening is associated with a substantial interval cancer rate in the region of 50 %, indicating a severe deficiency in sensitivity for cancer. Furthermore, as it is now well established that the majority of colorectal cancers arise from pre-existing adenomas, it is important for any colorectal screening programme to detect adenomas in order to reduce the incidence of the disease as well as the associated mortality. Although gFOBT does detect some adenomas, the randomised studies have not demonstrated a reduction in colorectal cancer incidence with the exception of the Minnesota Study that used rehydrated gFOBT resulting in a high positivity rate and a large number of colonoscopies. It should be borne in mind however, that the newer faecal immunochemical tests (FIT), which, unlike gFOBT, are specific for human haemoglobin, perform better in terms of both cancer and adenoma detection.

It is also of interest that recent scrutiny of the interval cancer data from the Scottish demonstration pilot has clearly demonstrated that gFOBT screening tends to under-detect cancers in women when compared with men. In addition, it is relatively insensitive for rectal cancer when compared with colon cancer. Analysis of quantitative FIT data in our laboratory as part of an evaluation of FIT as a first line test in Scotland, has shown that the mean faecal haemoglobin concentration in women is lower than that in men, and that the cutoff value required for women to give a 2% positivity rate (similar to that achieved by the gFOBT currently in use in the UK) is less than half that for men. Thus, for gender at least, FIT will have the same limitations as gFOBT.

In a recent randomised trial carried out in 14 UK centres, a single flexible sigmoidoscopy (FS) between the ages of 55 and 65 years has been shown to bring about a significant reduction in colorectal cancer mortality. In addition, and most importantly, after a period of four years a significant reduction in colorectal cancer incidence was observed, presumably as a result of the routine removal of adenomas at FS. Interestingly, the reduction in incidence was restricted to left-sided cancers despite the fact that total colonoscopy was carried out in all those with a significant index lesion found at FS (5% of the screened population). FS does not suffer from low specificity since false positives do not occur, and there is independent evidence that it is more sensitive than a single gFOBT or FIT. In addition, FS is ideally suited to detecting rectal cancers and adenomas, and it is unlikely that there would be a gender difference in the sensitivity.

This landmark study (henceforth referred to as the "UK FS trial") was, however, an efficacy study since it was carried out in a population who had already indicated an interest in participating and, as a result, the uptake in those randomised to FS was an impressive 71%. This, however, leaves significant questions surrounding the introduction of FS screening, as it is not clear how it would perform as a population screening tool. Extrapolation of the results of the FS trial to the general population would suggest an uptake in the region of around 30% and although it is not clear what the uptake of FS would be in the Scottish population, data from the Glasgow centre that participated in the FS indicate a likely uptake of 24%. This compares with an overall uptake of around 60% in the current Scottish Bowel Screening Programme based on gFOBT.

A population based randomised trial of FS from Norway achieved a participation rate of 67% but a randomised study from The Netherlands achieved an uptake of 32.4% for FS compared with 49.5% and 61.5% for gFOBT and FIT respectively. In addition, there is evidence that participants perceive the personal burden of FS to be greater than that of either type of faecal testing. On the other hand, a study from Italy found a similar participation rate or FIT and FS, although both were low at 32% of those invited. Two small studies conducted in the London area observed an uptake of screening FS of around 50% but a similar study carried out in Tayside, Scotland achieved an uptake of only 24%. It is not clear why there should be such discrepancies in uptake of FS, but both cultural issues and differences in levels of deprivation are likely to be important.

The randomised study from The Netherlands demonstrated that the diagnostic yield of advanced neoplasia (cancers and significant adenomas) per 100 invitees was greater for FS than for either of the faecal tests suggesting that the overall performance of FS may be better than faecal testing despite a lower participation rate. This introduces an important ethical dimension; namely, whether or not it is acceptable to use a population screening tool that reaches a relatively small proportion of the population rather than a test that is associated with a higher participation rate but has an overall poorer performance in terms of disease detection. This is further complicated by the adverse effect of deprivation on uptake of screening. It is known that, in Scotland, the difference in uptake of gFOBT population screening between the most deprived and the least deprived quintile is around 20%. The effect of deprivation on uptake of FS population screening is not known, although in the UK FS trial there was a 16% difference in intention to participate and a 20% difference in actual uptake in those invited between the most and least deprived quartiles in Glasgow.

In a recent re-appraisal of the options for colorectal cancer screening commissioned by the UK National Screening Committee, and based on the UK FS trial, data from the first two rounds of the English Bowel Screening Programme and data on the sensitivity and specificity of FIT, modelling has suggested that a single FS would perform better than biennial gFOBT and that FS at age 62 results in the greatest reduction in CRC incidence, CRC mortality and CRC treatment costs, whereas FS at age 54 results in the greatest gain in life years and QALYs. In addition it was suggested that biennial FIT may outperform both biennial gFOBT and one off FS.

As result, FS screening has been introduced into England for all at the age of 55. Thus it is offered 5 years before gFOBT screening starts, as this is offered between the ages of 60 and 74. In Scotland, however, the age range for gFOBT screening is 50 to 74, and the main issue surrounding the introduction of FS screening in Scotland is that there is no information regarding the utility of FS in a population that has already been exposed to FOBT screening.

Nevertheless, given the high degree of efficacy of FS screening, particularly in terms of disease prevention via adenoma detection, and the relatively higher participation associated with gFOBT screening and its potential to detect proximal cancers, it is hypothesised that offering a combination of both approaches would provide an enhanced screening algorithm that would be associated with better outcomes than either modality alone. In order to test this hypothesis and answer some key unresolved questions around FS, it is necessary to carry out a pilot of FS screening integrated into the current faecal test-based Scottish Screening Programme, and to maximise the information from this pilot it is proposed to carry it out as a random evaluation. It is also proposed that FS is offered at around the age of 60, as this appears to be the age at which adenoma prevalence peaks, and therefore the age at which adenoma detection and removal is likely to confer the maximum benefit. There is also evidence from the gFOBT pilot that 80% of interval cancers are diagnosed over the age of 60.

As the Scottish Bowel Screening Programme offers gFOBT from the age of 50, and as screening started in Grampian, Tayside and Fife in 2000 as part of the UK demonstration screening pilot, carrying out a study in these areas will demonstrate whether or not FS adds value to a mature biennial FOBT screening programme. Further evaluation in Greater Glasgow will test FS in a challenging Health Board with areas of high urban deprivation.

We will seek to establish the value and feasibility of flexible sigmoidoscopy in populations which have been exposed to gFOBT screening for colorectal cancer.

In this way it will be possible to estimate the added value of adding FS to the FOBT programme. This will inform the structure of the Scottish Bowel Screening Programme and provide information that will have international implications.

It will also be possible to estimate the practicalities of introducing flexible sigmoidoscopy into the Scottish population against a background of ongoing gFOBT screening.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for colorectal screening

Exclusion Criteria:

* Absence of colon

Ages: 59 Years to 61 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 4567 (Actual)
Dates: Start 2014-06; Primary Completion 2016-05 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Number of colorectal cancers or adenomas diagnosed | Within duration of study - two years
  Pathology report of lesion removed at flexible sigmoidoscopy or subsequent colonoscopy

SECONDARY OUTCOMES:
Number of invited individuals undergoing flexible sigmoidoscopy | Within duration of study - two years
  Record of whether or not the flexible sigmoidoscopy had been carried out

CONTACTS AND LOCATIONS:
Overall Officials: Robert JC Steele, MD, Principal Investigator — University of Dundee
Locations (1):
- NHS Tayside, Dundee, Scotland, United Kingdom

REFERENCES:
- [Background] Benson VS, Patnick J, Davies AK, Nadel MR, Smith RA, Atkin WS; International Colorectal Cancer Screening Network. Colorectal cancer screening: a comparison of 35 initiatives in 17 countries. Int J Cancer. 2008 Mar 15;122(6):1357-67. doi: 10.1002/ijc.23273. PMID 18033685
- [Background] Hewitson P, Glasziou P, Watson E, Towler B, Irwig L. Cochrane systematic review of colorectal cancer screening using the fecal occult blood test (hemoccult): an update. Am J Gastroenterol. 2008 Jun;103(6):1541-9. doi: 10.1111/j.1572-0241.2008.01875.x. Epub 2008 May 13. PMID 18479499
- [Background] Hardcastle JD, Chamberlain JO, Robinson MH, Moss SM, Amar SS, Balfour TW, James PD, Mangham CM. Randomised controlled trial of faecal-occult-blood screening for colorectal cancer. Lancet. 1996 Nov 30;348(9040):1472-7. doi: 10.1016/S0140-6736(96)03386-7. PMID 8942775
- [Background] Kronborg O, Fenger C, Olsen J, Jorgensen OD, Sondergaard O. Randomised study of screening for colorectal cancer with faecal-occult-blood test. Lancet. 1996 Nov 30;348(9040):1467-71. doi: 10.1016/S0140-6736(96)03430-7. PMID 8942774
- [Background] Lindholm E, Brevinge H, Haglind E. Survival benefit in a randomized clinical trial of faecal occult blood screening for colorectal cancer. Br J Surg. 2008 Aug;95(8):1029-36. doi: 10.1002/bjs.6136. PMID 18563785
- [Background] Steele RJ, McClements PL, Libby G, Black R, Morton C, Birrell J, Mowat NA, Wilson JA, Kenicer M, Carey FA, Fraser CG. Results from the first three rounds of the Scottish demonstration pilot of FOBT screening for colorectal cancer. Gut. 2009 Apr;58(4):530-5. doi: 10.1136/gut.2008.162883. Epub 2008 Nov 26. PMID 19036949
- [Background] Leslie A, Carey FA, Pratt NR, Steele RJ. The colorectal adenoma-carcinoma sequence. Br J Surg. 2002 Jul;89(7):845-60. doi: 10.1046/j.1365-2168.2002.02120.x. PMID 12081733
- [Background] Mandel JS, Bond JH, Church TR, Snover DC, Bradley GM, Schuman LM, Ederer F. Reducing mortality from colorectal cancer by screening for fecal occult blood. Minnesota Colon Cancer Control Study. N Engl J Med. 1993 May 13;328(19):1365-71. doi: 10.1056/NEJM199305133281901. PMID 8474513
- [Background] van Rossum LG, van Rijn AF, Laheij RJ, van Oijen MG, Fockens P, van Krieken HH, Verbeek AL, Jansen JB, Dekker E. Random comparison of guaiac and immunochemical fecal occult blood tests for colorectal cancer in a screening population. Gastroenterology. 2008 Jul;135(1):82-90. doi: 10.1053/j.gastro.2008.03.040. Epub 2008 Mar 25. PMID 18482589
- [Background] Steele RJ, McClements P, Watling C, Libby G, Weller D, Brewster DH, Black R, Carey FA, Fraser CG. Interval cancers in a FOBT-based colorectal cancer population screening programme: implications for stage, gender and tumour site. Gut. 2012 Apr;61(4):576-81. doi: 10.1136/gutjnl-2011-300535. Epub 2011 Sep 19. PMID 21930729
- [Background] McDonald PJ, Strachan JA, Digby J, Steele RJ, Fraser CG. Faecal haemoglobin concentrations by gender and age: implications for population-based screening for colorectal cancer. Clin Chem Lab Med. 2011 Dec 7;50(5):935-40. doi: 10.1515/CCLM.2011.815. PMID 22149740
- [Background] Atkin WS, Edwards R, Kralj-Hans I, Wooldrage K, Hart AR, Northover JM, Parkin DM, Wardle J, Duffy SW, Cuzick J; UK Flexible Sigmoidoscopy Trial Investigators. Once-only flexible sigmoidoscopy screening in prevention of colorectal cancer: a multicentre randomised controlled trial. Lancet. 2010 May 8;375(9726):1624-33. doi: 10.1016/S0140-6736(10)60551-X. Epub 2010 Apr 27. PMID 20430429
- [Background] Hol L, de Jonge V, van Leerdam ME, van Ballegooijen M, Looman CW, van Vuuren AJ, Reijerink JC, Habbema JD, Essink-Bot ML, Kuipers EJ. Screening for colorectal cancer: comparison of perceived test burden of guaiac-based faecal occult blood test, faecal immunochemical test and flexible sigmoidoscopy. Eur J Cancer. 2010 Jul;46(11):2059-66. doi: 10.1016/j.ejca.2010.03.022. Epub 2010 Jun 4. PMID 20621736
- [Background] McCaffery K, Wardle J, Nadel M, Atkin W. Socioeconomic variation in participation in colorectal cancer screening. J Med Screen. 2002;9(3):104-8. doi: 10.1136/jms.9.3.104. PMID 12370320
- [Background] Hoff G, Grotmol T, Skovlund E, Bretthauer M; Norwegian Colorectal Cancer Prevention Study Group. Risk of colorectal cancer seven years after flexible sigmoidoscopy screening: randomised controlled trial. BMJ. 2009 May 29;338:b1846. doi: 10.1136/bmj.b1846. PMID 19483252
- [Background] Hol L, van Leerdam ME, van Ballegooijen M, van Vuuren AJ, van Dekken H, Reijerink JC, van der Togt AC, Habbema JD, Kuipers EJ. Screening for colorectal cancer: randomised trial comparing guaiac-based and immunochemical faecal occult blood testing and flexible sigmoidoscopy. Gut. 2010 Jan;59(1):62-8. doi: 10.1136/gut.2009.177089. PMID 19671542
- [Background] Segnan N, Senore C, Andreoni B, Azzoni A, Bisanti L, Cardelli A, Castiglione G, Crosta C, Ederle A, Fantin A, Ferrari A, Fracchia M, Ferrero F, Gasperoni S, Recchia S, Risio M, Rubeca T, Saracco G, Zappa M; SCORE3 Working Group-Italy. Comparing attendance and detection rate of colonoscopy with sigmoidoscopy and FIT for colorectal cancer screening. Gastroenterology. 2007 Jun;132(7):2304-12. doi: 10.1053/j.gastro.2007.03.030. Epub 2007 Mar 21. PMID 17570205
- [Background] Verne JE, Aubrey R, Love SB, Talbot IC, Northover JM. Population based randomized study of uptake and yield of screening by flexible sigmoidoscopy compared with screening by faecal occult blood testing. BMJ. 1998 Jul 18;317(7152):182-5. doi: 10.1136/bmj.317.7152.182. PMID 9665902
- [Background] Robb K, Power E, Kralj-Hans I, Edwards R, Vance M, Atkin W, Wardle J. Flexible sigmoidoscopy screening for colorectal cancer: uptake in a population-based pilot programme. J Med Screen. 2010;17(2):75-8. doi: 10.1258/jms.2010.010055. PMID 20660435
- [Background] Gray M, Pennington CR. Screening sigmoidoscopy: a randomised trial of invitation style. Health Bull (Edinb). 2000 Mar;58(2):137-40. PMID 12813842
- [Background] Steele RJ, Kostourou I, McClements P, Watling C, Libby G, Weller D, Brewster DH, Black R, Carey FA, Fraser C. Effect of gender, age and deprivation on key performance indicators in a FOBT-based colorectal screening programme. J Med Screen. 2010;17(2):68-74. doi: 10.1258/jms.2010.009120. PMID 20660434
- [Background] Atkin WS, Cuzick J, Northover JM, Whynes DK. Prevention of colorectal cancer by once-only sigmoidoscopy. Lancet. 1993 Mar 20;341(8847):736-40. doi: 10.1016/0140-6736(93)90499-7. PMID 8095636